CLINICAL TRIAL: NCT00538434
Title: An Efficacy and Safety Study of Reslizumab (CTx55700) in the Treatment of Eosinophilic Esophagitis in Subjects Aged 5 to 18 Years
Brief Title: Efficacy and Safety Study of Reslizumab to Treat Eosinophilic Esophagitis in Subjects Aged 5 to 18 Years
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ception Therapeutics (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Res-05-0002
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Results first posted 2016-09-02 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-07

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis; GERD; EE; Reslizumab; IL-5; Interleukin-5; Cinquil
MeSH Terms: conditions — Eosinophilic Esophagitis; Gastroesophageal Reflux | interventions — reslizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Reslizumab 1 mg/kg (Experimental): reslizumab 1 mg/kg intravenous (IV) on Day 0 of each 28-day (+/-7 days) cycle, for up to 4 cycles
  Interventions: Biological: Reslizumab
- Reslizumab 2 mg/kg (Experimental): reslizumab 2 mg/kg IV on Day 0 of each 28-day (+/-7 days) cycle, for up to 4 cycles
  Interventions: Biological: Reslizumab
- Reslizumab 3 mg/kg (Experimental): reslizumab 3 mg/kg IV on Day 0 of each 28-day (+/-7 days) cycle, for up to 4 cycles
  Interventions: Biological: Reslizumab
- Placebo (Placebo Comparator): saline placebo IV on Day 0 of each 28-day (+/-7 days) cycle, for up to 4 cycles
  Interventions: Other: Saline

INTERVENTIONS:
Biological: Reslizumab
  Other Names: CTx55700; Cinquil™; CEP-38072
  Arms: Reslizumab 1 mg/kg; Reslizumab 2 mg/kg; Reslizumab 3 mg/kg
Other: Saline
  Arms: Placebo

SUMMARY:
This trial will study three doses of reslizumab versus placebo in children with eosinophilic esophagitis (EE). The objectives of the trial will be to study the effectiveness of reslizumab in improving the clinical signs and symptoms and reducing esophageal eosinophils as well as assessing the safety profile compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent obtained
* male or female patients aged 5 to 18 years at time of screening
* of non-childbearing potential, of childbearing potential and willing to use specific barrier methods outlined in the protocol
* confirmed active EE (at Screening or within six weeks prior to Baseline Visit) as defined by esophageal mucosal eosinophils greater than or equal to 24 per high power field (hpf; 400X magnification)
* within the week prior to dosing, patient has one of the following symptoms of moderate (or worse) severity: vomiting, regurgitation (acid taste or feeling material movement upward), abdominal, chest pain/heartburn (burning or pain behind the sternum), or difficulty swallowing
* been on a therapeutic dose of proton pump inhibitors (PPIs; with or without histamine H2 receptor antagonists)for at least four weeks without resolution of symptoms, or by negative pH probe (with or without having failed a course of PPIs)

Exclusion Criteria:

* another disorder that causes esophageal eosinophilia (e.g., hypereosinophilic syndrome [HES],Churg Strauss vasculitis, eosinophilic gastroenteritis [EG], or a parasitic infection)
* history of abnormal gastric or duodenal biopsy or documented gastrointestinal [GI] disorders (e.g., celiac disease, Crohn's disease or Helicobacter pylori infection)
* history of the following GI surgeries: fundoplication, gastric surgery or surgery for intestinal atresia
* use of systemic immunosuppressive or immunomodulating agents (anti-immunoglobulin E [IgE] monoclinal antibody [mAb], methotrexate, cyclosporin, interferon alpha [α], or anti tumor necrosis factor [TNF] mAb) within six months prior to study entry
* received attenuated live attenuated vaccines (e.g., measles, mumps, rubella [MMR], bacillus Calmette-Guerin [BCG], varicella, FluMist or polio) within three months prior to study entry
* use of swallowed inhaled corticosteroids for the treatment of EE within one month prior to study entry. Note: Inhaled and nasal corticosteroids for the treatment of asthma and allergies, respectively, are permitted provided that the dose remains the same during the study
* a stricture on endoscopy that prevents passage of the endoscope
* participation in any investigational drug or device study within 30 days prior to study entry
* female subjects who are pregnant or nursing
* concurrent infection or disease that may preclude assessment of EE
* concurrent immunodeficiency (human immunodeficiency [HIV], or acquired immunodeficiency syndrome [AIDS] or congenital immunodeficiency)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 227 (Actual)
Dates: Start 2008-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, MD, Study Director — Cephalon (Ception)
Locations (37):
- United States (34):
  - The Children's Hospital of Alabama, Birmingham, Alabama
  - University of Arizona Dept. of Pediatrics, Tucson, Arizona
  - Arkansas Children's Hospital/University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Hospital- Pediatric Gastroenterology, Hayward, California
  - Children'S Hospital of Orange County Pediatric Subspecialty Faculty Division of Allergy and Asthma, Orange, California
  - Pediatric Allergy/Immunology, Palo Alto, California
  - Children's Hospital of San Diego, San Diego, California
  - Denver Childrens At Aurora, Colorado, Aurora, Colorado
  - 1st Allergy and Clinical Research Center, Centennial, Colorado
  - Thomas Jefferson University Medical College, Wilmington, Delaware
  - Children's Center for Digestive Health Care, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Children'S Memorial Hospital Division of Gastroenterology Hepatology & Nutrition, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Tuft's Floating Hospital, Boston, Massachusetts
  - Minnesota Gastroenterology, Plymouth, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Creighton University Medical Center, Omaha, Nebraska
  - Las Vegas Pediatric Gastroenterology Associates, Las Vegas, Nevada
  - South Jersey Pediatric Gastroenterology, Mays Landing, New Jersey
  - Mount Sinai School of Medicine, Pediatrics, New York, New York
  - State University of New York (SUNY), Syracuse, New York
  - Center for Digestive Allergic and Immunologic Diseases, Williamsville, New York
  - Pediatric Allergy and Immunology of Duke Medical Center, Durham, North Carolina
  - Cincinnati Children's, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - University of Texas Southwest Medical Center, Dallas, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Carilion Medical Center for Children, Roanoke, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - Pediatric Allergy and Immunology, Edmonton, Alberta
  - Pediatric Allergy & Immunology, Edmonton, Alberta
  - University of Montreal, Montreal, Quebec

REFERENCES:
- [Result] Spergel JM, Rothenberg ME, Collins MH, Furuta GT, Markowitz JE, Fuchs G 3rd, O'Gorman MA, Abonia JP, Young J, Henkel T, Wilkins HJ, Liacouras CA. Reslizumab in children and adolescents with eosinophilic esophagitis: results of a double-blind, randomized, placebo-controlled trial. J Allergy Clin Immunol. 2012 Feb;129(2):456-63, 463.e1-3. doi: 10.1016/j.jaci.2011.11.044. Epub 2011 Dec 28. PMID 22206777

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reslizumab 1 mg/kg | Reslizumab 2 mg/kg | Reslizumab 3 mg/kg | Placebo
Started | 56 | 57 | 57 | 57
Intent-to-treat (ITT) Population | 55 (1 participant was randomized but not treated) | 57 | 57 | 57
Completed | 47 (Completed all scheduled study visits) | 46 (Completed all scheduled study visits) | 50 (Completed all scheduled study visits) | 51 (Completed all scheduled study visits)
Not Completed | 9 | 11 | 7 | 6

BASELINE CHARACTERISTICS:
Population: ITT population: all randomized participants who received any amount of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Reslizumab 1 mg/kg | Reslizumab 2 mg/kg | Reslizumab 3 mg/kg | Placebo | Total
Number analyzed (Participants) | 55 | 57 | 57 | 57 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.3 (3.83) | 11.8 (3.82) | 11.5 (4.04) | 11.9 (4.17) | 11.9 (3.95)
Age, Customized [Number; unit: participants]
  5 to < 12 years | 21 | 26 | 27 | 25 | 99
  12 to < 19 years | 34 | 31 | 30 | 32 | 127
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 12 | 13 | 54
  Male | 41 | 42 | 45 | 44 | 172

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline to End of Treatment in Peak Esophageal Eosinophil (EE) Levels
Description: Participants underwent esophagogastroduodenoscopy (EGD) with biopsy (2 biopsies each at proximal and distal esophageal locations, plus any inflamed or abnormal areas) per standard clinical practice for the determination of esophageal eosinophils.
Time Frame: Baseline, End of Treatment (up to 15 weeks [+/- 4 days])
Population: ITT population: all randomized participants who received any amount of study drug.
Measure: Mean (Standard Deviation); unit: percentage change in eosinophils/hpf
Arm/Group | Reslizumab 1 mg/kg | Reslizumab 2 mg/kg | Reslizumab 3 mg/kg | Placebo
Number analyzed (Participants) | 55 | 57 | 57 | 57
percentage change in eosinophils/hpf | -37.60 (70.86) | -58.27 (35.45) | -56.46 (34.82) | 11.50 (91.42)
Statistical Analysis 1: Comparison: Reslizumab 1 mg/kg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; adjustment for stratification factor and for variable at Baseline; Adjusted mean difference = -52.78, 95% CI 2-sided [-75.24 to -30.32], Standard Error of Mean 11.40
Statistical Analysis 2: Comparison: Reslizumab 2 mg/kg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; adjustment for stratification factor and for variable at Baseline; Adjusted mean difference = -73.03, 95% CI 2-sided [-95.28 to -50.78], Standard Error of Mean 11.29
Statistical Analysis 3: Comparison: Reslizumab 3 mg/kg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; adjustment for stratification factor and for variable at Baseline; Adjusted mean difference = -64.69, 95% CI 2-sided [-86.93 to -42.45], Standard Error of Mean 11.28

2. Primary Outcome: Mean Change From Baseline in Physician's Esophageal Eosinophil (EE) Global Assessment At The End-of-Treatment Visit (or at Early Withdrawal)
Description: The investigator completed the Physician's EE Global Assessment based upon the participant's reporting of symptoms, weight, dietary status, and overall well-being. The assessment rated severity on a five-point scale (0=none to 4=very severe), taking into account physical findings, vital signs, the Subject's Predominant EE Symptom Assessment, the subject's diary data, and dietary questions. The Subject's Predominant EE Symptom was the EE symptom (vomiting/regurgitation, abdominal/chest pain, or dysphagia) that had the greatest negative impact on the subject based on patient diary data as of the baseline visit.
  The full range for change from baseline values is -4 (very severe at baseline, none at end of study) to 4 (none at baseline, severe at end of study). Negative change from baseline scores in the Physician's EE Global Assessment indicate improvement in EE status.
Time Frame: Baseline (Day 1, pre-treatment), End of Treatment (Week 15, 3 weeks [± 4 days] after the last dose of study drug, or at early withdrawal)
Population: ITT population: all randomized participants who received any amount of study drug with both a baseline and an End of Treatment assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Reslizumab 1 mg/kg | Reslizumab 2 mg/kg | Reslizumab 3 mg/kg | Placebo
Number analyzed (Participants) | 55 | 57 | 57 | 57
units on a scale | -0.85 (NA) — Study documentation from an acquired company does not contain the measure of dispersion. | -1.02 (NA) — Study documentation from an acquired company does not contain the measure of dispersion. | -1.12 (NA) — Study documentation from an acquired company does not contain the measure of dispersion. | -1.14 (NA) — Study documentation from an acquired company does not contain the measure of dispersion.
Statistical Analysis 1: Comparison: Reslizumab 1 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.0313, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Reslizumab 2 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.5793, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Reslizumab 3 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.4905, Cochran-Mantel-Haenszel

3. Secondary Outcome: Mean Change From Baseline to End of Treatment in EE Predominant Symptom Assessment
Description: Participants rated the severity of each EE symptom (vomiting/regurgitation, abdominal/chest pain, and dysphagia) based on the previous week's daily diary as none (=0), mild, moderate, severe, or very severe (=4). The predominant symptom was selected at the baseline visit and remained the same throughout the trial. The predominant symptom was defined as the EE symptom that had the greatest negative impact on the participant. The full range for change from baseline values is -4 (very severe at baseline, none at end of study) to 4 (none at baseline, severe at end of study). Negative change from baseline scores in the Patient's EE Predominant Symptom Assessment indicate improvement in the selected symptom.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Reslizumab 1 mg/kg | Reslizumab 2 mg/kg | Reslizumab 3 mg/kg | Placebo
Number analyzed (Participants) | 54 | 56 | 57 | 55
units on a scale | -0.94 (NA) — Study documentation from an acquired company does not contain the measure of dispersion. | -1.20 (NA) — Study documentation from an acquired company does not contain the measure of dispersion. | -1.28 (NA) — Study documentation from an acquired company does not contain the measure of dispersion. | -1.44 (NA) — Study documentation from an acquired company does not contain the measure of dispersion.
Statistical Analysis 1: Comparison: Reslizumab 1 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.0062, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Reslizumab 2 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.0943, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Reslizumab 3 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.2955, Cochran-Mantel-Haenszel

4. Secondary Outcome: Mean Percent Change From Baseline to End of Treatment in the Child Health Questionnaire (CHQ)
Description: CHQ is a quality-of-life (QoL), observer-rated (the parent in this study) instrument designed to assess the general health and well-being of pediatric subjects aged 5 to 18 years. The instrument comprises 50 items that cover 14 unique physical and psychological concepts. Each item was scored separately following different scales and timeframes for response. Proprietary scoring algorithms are used. This outcome reports the two CHQ Summary Scores (Physical Summary Score and the Psychosocial Summary Scores) which are indexed to a 0 (poorest quality of life) to 100 (best quality of life) scores. The two summary scores are subsequently combined (via proprietary algorithm) to create the Global Health Summary Score (also on a 0-100 scale). Percent change from baseline values range from 100% (poorest QoL at baseline, best QoL at end of treatment) to -100% (best QoL at baseline, poorest QoL at end of treatment). Higher percent change from baseline values indicate improved QoL.
Time Frame: Baseline, End of Treatment (up to 15 weeks +/- 4 days)
Population: ITT population: all randomized participants who received any amount of study drug with both a baseline and an End of Treatment assessment; n=number of participants with a response in the given category.
Measure: Mean (Standard Deviation); unit: percentage change in score
Groups:
- Reslizumab 2 mg/kg: reslizumab 2 mg/kg intravenous (IV) on Day 0 of each 28-day (+/-7 days) cycle, for up to 4 cycles
Arm/Group | Reslizumab 1 mg/kg | Reslizumab 2 mg/kg | Reslizumab 3 mg/kg | Placebo
Number analyzed (Participants) | 55 | 57 | 57 | 57
percentage change in score
  Physical Summary Score; n=49, 52, 53, 57 | 11.2 (NA) — Study documentation from an acquired company does not contain the measure of dispersion. | 18.6 (NA) — Study documentation from an acquired company does not contain the measure of dispersion. | 18.5 (NA) — Study documentation from an acquired company does not contain the measure of dispersion. | 11.8 (NA) — Study documentation from an acquired company does not contain the measure of dispersion.
  Psychosocial Summary Score; n=51, 52, 53, 55 | 5.0 (NA) — Study documentation from an acquired company does not contain the measure of dispersion. | 12.2 (NA) — Study documentation from an acquired company does not contain the measure of dispersion. | 14.1 (NA) — Study documentation from an acquired company does not contain the measure of dispersion. | 10.1 (NA) — Study documentation from an acquired company does not contain the measure of dispersion.
  Global Health Summary Score; n=50, 54, 54, 55 | 10.2 (NA) — Study documentation from an acquired company does not contain the measure of dispersion. | 15.5 (NA) — Study documentation from an acquired company does not contain the measure of dispersion. | 10.3 (NA) — Study documentation from an acquired company does not contain the measure of dispersion. | 9.7 (NA) — Study documentation from an acquired company does not contain the measure of dispersion.
Statistical Analysis 1: Comparison: Reslizumab 1 mg/kg vs Placebo; Physical Summary Score; Test type: Superiority or Other; p = 0.4644, ANCOVA — Analyzed using analysis of covariance with adjustment for stratification factor and for variable at baseline; Adjusted mean difference = -4.75, 95% CI 2-sided [-17.53 to 8.03], Standard Error of Mean 6.48 — Comparison of least square means provides the difference (of individual change scores) between each reslizumab dose group and placebo
Statistical Analysis 2: Comparison: Reslizumab 2 mg/kg vs Placebo; Physical Summary Score; Test type: Superiority or Other; p = 0.8196, ANCOVA — Analyzed using analysis of covariance with adjustment for stratification factor and for variable at baseline; Adjusted mean difference = -1.47, 95% CI 2-sided [-14.17 to 11.23], Standard Error of Mean 6.44 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Reslizumab 3 mg/kg vs Placebo; Physical Summary Score; Test type: Superiority or Other; p = 0.8306, ANCOVA — Analyzed using analysis of covariance with adjustment for stratification factor and for variable at baseline; Adjusted mean difference = 1.36, 95% CI 2-sided [-11.19 to 13.91], Standard Error of Mean 6.36 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Reslizumab 1 mg/kg vs Placebo; Psychosocial Summary Score; Test type: Superiority or Other; p = 0.1459, ANCOVA — Analyzed using analysis of covariance with adjustment for stratification factor and for variable at baseline; Adjusted mean difference = -6.38, 95% CI 2-sided [-15.01 to 2.24], Standard Error of Mean 4.37 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Reslizumab 2 mg/kg vs Placebo; Psychosocial Summary Score; Test type: Superiority or Other; p = 0.4375, ANCOVA — Analyzed using analysis of covariance with adjustment for stratification factor and for variable at baseline; Adjusted mean difference = -3.41, 95% CI 2-sided [-12.05 to 5.23], Standard Error of Mean 4.38 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Reslizumab 3 mg/kg vs Placebo; Psychosocial Summary Score; Test type: Superiority or Other; p = 0.9217, ANCOVA — Analyzed using analysis of covariance with adjustment for stratification factor and for variable at baseline; Adjusted mean difference = -0.43, 95% CI 2-sided [-9.00 to 8.15], Standard Error of Mean 4.35 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: Reslizumab 1 mg/kg vs Placebo; Global Health Score; Test type: Superiority or Other; p = 0.8412, ANCOVA — Analyzed using analysis of covariance with adjustment for stratification factor and for variable at baseline; Adjusted mean difference = -1.57, 95% CI 2-sided [-16.98 to 13.85], Standard Error of Mean 7.82 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: Reslizumab 2 mg/kg vs Placebo; Global Health Score; Test type: Superiority or Other; p = 0.4794, ANCOVA — Analyzed using analysis of covariance with adjustment for stratification factor and for variable at baseline; Adjusted mean difference = -5.54, 95% CI 2-sided [-20.94 to 9.87], Standard Error of Mean 7.81 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 9: Comparison: Reslizumab 3 mg/kg vs Placebo; Global Health Score; Test type: Superiority or Other; p = 0.8906, ANCOVA — Analyzed using analysis of covariance with adjustment for stratification factor and for variable at baseline; Adjusted mean difference = -1.06, 95% CI 2-sided [-16.16 to 14.06], Standard Error of Mean 7.66 — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: Baseline through Safety Follow-up (Week 16)
Arm/Group | Reslizumab 1 mg/kg | Reslizumab 2 mg/kg | Reslizumab 3 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/55 | 1/57 | 1/57 | 2/57
Other Adverse Events (participants affected / at risk) | 38/55 | 29/57 | 39/57 | 40/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reslizumab 1 mg/kg (N=55) | Reslizumab 2 mg/kg (N=57) | Reslizumab 3 mg/kg (N=57) | Placebo (N=57)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reslizumab 1 mg/kg (N=55) | Reslizumab 2 mg/kg (N=57) | Reslizumab 3 mg/kg (N=57) | Placebo (N=57)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 (7) | 0 (0) | 3 (3) | 2 (2)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 (4) | 2 (2) | 4 (5) | 5 (8)
DIARRHOEA (Gastrointestinal disorders) | 4 (4) | 3 (3) | 0 (0) | 5 (8)
NAUSEA (Gastrointestinal disorders) | 6 (6) | 2 (2) | 4 (4) | 3 (3)
VOMITING (Gastrointestinal disorders) | 2 (2) | 2 (3) | 2 (4) | 5 (5)
CHEST PAIN (General disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
FATIGUE (General disorders) | 5 (7) | 2 (6) | 3 (6) | 1 (1)
PYREXIA (General disorders) | 4 (5) | 2 (2) | 3 (4) | 6 (8)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 2 (2) | 0 (0) | 4 (4) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 7 (8)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 3 (3)
SINUSITIS (Infections and infestations) | 5 (5) | 1 (1) | 5 (6) | 4 (4)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 (5) | 4 (4) | 6 (6) | 5 (6)
VIRAL INFECTION (Infections and infestations) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
PROTEIN URINE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
RED BLOOD CELLS URINE POSITIVE (Investigations) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
URINARY CASTS (Investigations) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
URINE OXALATE INCREASED (Investigations) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
WHITE BLOOD CELLS URINE POSITIVE (Investigations) | 4 (7) | 0 (0) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 2 (3) | 1 (1) | 6 (7) | 1 (2)
HEADACHE (Nervous system disorders) | 8 (9) | 6 (7) | 12 (15) | 7 (7)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (7) | 6 (7) | 6 (6)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 3 (3) | 4 (4) | 8 (9)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 4 (5) | 9 (12)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 0 (0) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.